CLINICAL TRIAL: NCT05377021
Title: A New Approach Intended for the Examination of "Diet" and "Diet and Exercise Combination" Interventions in Obese Women With Polycystic Ovary Syndrome
Brief Title: Lifestyle Change in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Hülya Özberk, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DokuzEU123
Record Dates: First submitted 2022-05-09; First posted 2022-05-17 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2022-05

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Intervention Model Description: A prospective and randomized comparison
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Diet" group (Active Comparator)
  Interventions: Behavioral: Lifestyle change
- "Diet and exercise combination" group (Experimental)
  Interventions: Behavioral: Lifestyle change

INTERVENTIONS:
Behavioral: Lifestyle change — In the project, 33 women in the first group will receive "diet" intervention for 12 weeks, and 33 women in the second group will receive "diet and exercise combination" intervention.
  Other Names: Lifestyle change in women with polycystic ovary syndrome

SUMMARY:
This project aims to compare "diet" and "diet and exercise combination" interventions in obese women with polycystic ovary syndrome.

This project will be carried out in the Dokuz Eylül University Research and Application Hospital gynecology outpatient clinic between June 1, 2022 and June 1, 2024. The purpose of the project will be explained to women who meet the sampling criteria, and their informed consent will be obtained. A prospective and randomized comparison of "diet" and "diet and exercise combination" interventions, which are among the first-line treatment lifestyle changes recommended for PCOS, will be done. In the project, 33 women in the first group will receive "diet" intervention for 12 weeks, and 33 women in the second group will receive "diet and exercise combination" intervention. "Descriptive Characteristics Form" will be filled in for both groups, then at the beginning and at the end of the project, routine ultrasonography and laboratory test parameters for PCOS diagnosis criteria and menstrual cycle characteristics will be recorded, hirsutism score, alopecia score and acne level will be evaluated, the Utian Quality of Life Scale, Body Appreciation Scale, and the Short Form of the Oxford Happiness Questionnaire will be filled out. Body composition analysis will be performed in both groups at the beginning of the project, in the fourth and eighth weeks, and personal dietary recommendations will be given. Kitchen scales will be given to both groups to adapt to dietary recommendations and a mobile nutrition application will be used to record their diets. Person-specific exercise recommendations will be given to the second group at the beginning of the project, in the fourth and eighth weeks. In addition, women will be informed with a guide to behavioral changes specific to PCOS, which will be prepared specific to their group. Exercise parameters will be recorded by giving the same mobile application. Mobile nutrition application data will be collected via e-mail in the fourth, eighth and twelfth weeks of the project.

ELIGIBILITY:
Inclusion Criteria:

* Being between 20-41 years old,
* Diagnosis of polycystic ovary syndrome,
* Having a secondary education or higher education,
* Having a body mass index of 30 and above,
* Volunteering to participate in the research

Exclusion Criteria:

* Having a psychiatric diagnosis,
* Using a contraceptive method containing hormones in the last three months,
* Presence of one or more of the etiologies of hyperprolactinemia, thyroid dysfunction, Cushing's syndrome, congenital adrenal hyperplasia and other hyperandrogenemia,
* Diagnosis of hypertension, Type 1 or Type 2 Diabetes Mellitus,
* Using one or more of the drug types such as antiandrogen, steroid, antidiabetic, ovulation induction agents in the last three months,
* Impairment of liver, kidney or heart functions,
* Limited physical exercise

Ages: 20 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
The smartwatch was evaluated as the primary outcome measure to assess the difference between the two groups. | 12 weeks
  Monthly average number of steps between groups
The mobile nutrition app was evaluated as the primary outcome measure to assess the difference between the two groups. | 12 weeks
  Average monthly calorie intake between groups
Changes in body mass index (BMI) of women with polycystic ovary syndrome | 12 weeks
  Changes in BMI will be evaluated using kg/m^2.

SECONDARY OUTCOMES:
Quality of life of women with polycystic ovary syndrome | 12 weeks
  Quality of life assessed by Utian Quality of Life Scale. This scale consists of five-point Likert type, 23 items and four sub-dimensions (health, emotional, sexual and occupational quality of life). The lowest score that can be obtained from the scale is 23, and the highest score is 115. An increase in the scale and sub-dimension scores indicates that the quality of life increases. The Cronbach Alpha coefficient of the scale is 0.88.
Satisfaction of women with polycystic ovary syndrome | 12 weeks
  Satisfaction assessed by Body Satisfaction Scale. This scale is five-point Likert type. It consists of two factors, general body satisfaction and investment in body image, and nine items. High scores from the scale reflect high body satisfaction. The Cronbach Alpha coefficient of the scale is 0.87.
The number of ovarian cysts | 12 weeks
  Ultrasound measurements 12 weeks later
The value of hirsutism among PCOS symptoms between the groups | 12 weeks
  Ferriman-Gallwey score (mFG) system was used for hirsutism.
The grade of alopecia among PCOS symptoms between the groups | 12 weeks
  the Ludwig classification system was used.
The value of acne among PCOS symptoms between the groups | 12 weeks
  The Global Acne Grading System was used.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylül University, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Available from the researcher upon request.